CLINICAL TRIAL: NCT07387822
Title: Effect of Individualized Versus Standardized Open-Lung Ventilation on Postoperative Pulmonary Complications in Thoracic Surgery: A Randomized Controlled Trial
Brief Title: Individualized Open Lung Ventilation and Postoperative Pulmonary Complications in Thoracic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Xinrui Yin, Doctor, Aerospace Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYin-Trial-2026-01-08
Record Dates: First submitted 2026-01-08; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pulmonary Complications (PPCs); One-lung Ventilation (OLV); Thoracic Surgery, Video Assisted
Keywords: Individualized Open Lung Ventilation; Driving Pressure; PEEP Titration; Lung Recruitment Maneuver; Lung Protective Ventilation; Video-Assisted Thoracic Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Lung-Protective Ventilation Group (Active Comparator)
  Interventions: Procedure: Standard Lung-Protective Ventilation
- Individualized Open Lung Ventilation Group (Experimental)
  Interventions: Procedure: Individualized Open Lung Ventilation

INTERVENTIONS:
Procedure: Standard Lung-Protective Ventilation — Standard lung-protective ventilation is applied during one-lung ventilation. Ventilation parameters include a tidal volume of 6 mL/kg predicted body weight and a fixed positive end-expiratory pressure (PEEP) of 5 cmH2O throughout one-lung ventilation. No routine recruitment maneuver is performed during one-lung ventilation. At the end of one-lung ventilation, a standardized lung recruitment maneuver is applied before resuming two-lung ventilation.
  Arms: Standard Lung-Protective Ventilation Group
Procedure: Individualized Open Lung Ventilation — Individualized open lung ventilation is applied during one-lung ventilation. Tidal volume is set at 4-6 mL/kg predicted body weight. After lung recruitment, a decremental PEEP trial is performed starting from 10 cmH2O, with PEEP reduced stepwise to identify the level associated with the lowest driving pressure. The selected PEEP is maintained throughout one-lung ventilation. A standardized lung recruitment maneuver is applied at the end of one-lung ventilation before resuming two-lung ventilation.
  Arms: Individualized Open Lung Ventilation Group

SUMMARY:
This prospective, single-center, randomized controlled trial aims to evaluate the efficacy of an intraoperative "Individualized Open Lung Ventilation" strategy compared to a standard lung-protective ventilation strategy in patients undergoing thoracic surgery.

One-lung ventilation (OLV) is essential for thoracic surgery but can cause lung injury. While standard care often uses fixed ventilation parameters, this study investigates whether personalizing Positive End-Expiratory Pressure (PEEP) to achieve the lowest driving pressure can reduce the incidence of postoperative pulmonary complications (PPCs) within 7 days after surgery.

DETAILED DESCRIPTION:
Background: Postoperative pulmonary complications (PPCs) are a major cause of morbidity following thoracic surgery. One-lung ventilation (OLV), while necessary for surgical exposure, induces ischemia-reperfusion injury and mechanical stress. Current standard lung-protective ventilation (LPV) strategies typically employ low tidal volumes with a fixed Positive End-Expiratory Pressure (PEEP). However, fixed parameters may not account for individual variations in lung compliance and mechanics. This study hypothesizes that an individualized open lung approach, guided by driving pressure, will optimize lung mechanics and reduce clinical complications.

Study Design: This is a prospective, randomized controlled trial conducted at Aerospace Center Hospital. Eligible patients aged 18-75 undergoing elective video-assisted thoracic surgery (VATS) with an expected OLV duration of >1 hour will be enrolled.

Intervention Groups: Participants are randomized (1:1) into two groups:

Control Group (Standard Strategy): Patients receive volume-controlled ventilation during OLV with a tidal volume of 6 mL/kg predicted body weight (PBW) and a fixed PEEP of 5 cmH2O. No routine lung recruitment maneuvers are performed.

Experimental Group (Individualized Strategy): Patients receive a tidal volume of 4-6 mL/kg PBW. Upon initiating OLV, a lung recruitment maneuver is performed (PEEP increased to 10 cmH2O). Subsequently, a decremental PEEP trial is conducted (starting at 10 cmH2O and decreasing by 1 cmH2O steps) to identify the optimal PEEP level that produces the lowest driving pressure. This optimal PEEP is maintained for the duration of OLV.

Outcomes: The primary outcome is the incidence of defined Postoperative Pulmonary Complications (PPCs) within 7 days post-surgery, including pneumonia, atelectasis, ARDS, respiratory failure, and re-intubation. Secondary outcomes include intraoperative respiratory mechanics (driving pressure, compliance, oxygenation index), length of hospital stay, and other system complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Body mass index between 18 and 30 kg/m².
* Scheduled for elective video-assisted thoracoscopic surgery (VATS).
* Expected duration of one-lung ventilation longer than 1 hour.
* Able to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Emergency surgery or reoperation.
* History of severe pulmonary disease, including chronic obstructive pulmonary disease, pulmonary fibrosis, severe emphysema, pulmonary bullae, pneumothorax, or uncontrolled asthma.
* History of heart failure or coronary artery disease.
* Previous thoracic surgery or mechanical ventilation within 1 month before surgery.
* Planned postoperative mechanical ventilation.
* Bilateral thoracic surgery.
* Participation in another interventional clinical trial.
* Conversion to open thoracotomy during surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications within 7 days | Within 7 days after surgery
  Postoperative pulmonary complications (PPCs) occurring within 7 days after surgery, defined according to pre-specified criteria, including pneumonia, atelectasis requiring therapeutic intervention, acute respiratory distress syndrome (ARDS), respiratory failure requiring noninvasive or invasive mechanical ventilation, reintubation, or mechanical ventilation lasting longer than 48 hours.

SECONDARY OUTCOMES:
Incidence of secondary postoperative pulmonary complications within 30 days | Within 30 days after surgery
  Secondary postoperative pulmonary complications occurring within 30 days after surgery, including mild atelectasis, pleural effusion, bronchospasm, prolonged air leak, and other pulmonary complications not meeting the criteria for primary postoperative pulmonary complications.
Intraoperative Driving Pressure | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  Driving pressure is calculated as the difference between Plateau Pressure and Positive End-Expiratory Pressure. Lower driving pressure indicates lung-protective ventilation. Assessments are performed at 5 predefined time points: T1 (TLV baseline after positioning), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Incidence of non-pulmonary postoperative complications | Within 30 days after surgery
  Postoperative non-pulmonary complications within 30 days after surgery, including cardiovascular, neurological, gastrointestinal, urinary, and wound-related complications.
Intraoperative Dynamic Compliance | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  Dynamic compliance is measured as Tidal Volume divided by (Peak Pressure - PEEP). Higher compliance suggests better lung mechanics. Data is collected at T1 (TLV baseline), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Intraoperative Peak Airway Pressure | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  The maximum pressure measured during the inspiratory phase of the mechanical ventilation cycle. Data is collected at 5 predefined time points: T1 (TLV baseline after positioning), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Arterial Oxygen Partial Pressure to Fractional Inspired Oxygen Ratio | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  Ratio of arterial oxygen partial pressure to fractional inspired oxygen, assessed by arterial blood gas analysis to evaluate oxygenation status. Assessments are performed at: T1 (TLV baseline), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Hospital Length of Stay | Participants will be followed for the duration of hospital stay, an average of 7-9 days.
  he total duration of hospital stay from admission to discharge.
Incidence of ICU Admission | From date of surgery until date of discharge, assessed up to 30 days
  Number of participants requiring admission to the Intensive Care Unit after surgery.
30-Day Mortality | 30 days post-surgery
  All-cause mortality occurring within 30 days after surgery.
Incidence of Intraoperative Hypotension | From the start of anesthesia induction until the end of surgery.
  Defined as a mean arterial pressure < 65 mmHg or a > 20% decrease from baseline requiring vasopressor support.
Incidence of Pneumothorax | Within 7 days after surgery.
  Occurrence of pneumothorax detected postoperatively.
Partial Pressure of Carbon Dioxide | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  PaCO2 levels measured by arterial blood gas analysis. Measurements correspond to 5 time points: T1 (TLV baseline), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Arterial pH | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  Acid-base status assessed by arterial blood gas analysis. Measurements correspond to 5 time points: T1 (TLV baseline), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Mean Arterial Pressure | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  Average blood pressure in an individual during a single cardiac cycle. Data is recorded at: T1 (TLV baseline), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).
Heart Rate | From the start of mechanical ventilation until 15 minutes after the restoration of two-lung ventilation.
  Frequency of the cardiac cycle measured in beats per minute. Data is recorded at: T1 (TLV baseline), T2 (OLV 30 minutes), T3 (OLV 60 minutes), T4 (during resection), and T5 (within 15 minutes of TLV restoration).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangli Zheng, Principal Investigator — Aerospace Center Hospital
Locations (1):
- Aerospace Center Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Caplan JP, Chang G. Refeeding syndrome as an iatrogenic cause of delirium: a retrospective pilot study. Psychosomatics. 2010 Sep-Oct;51(5):419-24. doi: 10.1176/appi.psy.51.5.419. PMID 20833941
- [Result] Dulski J, Middlebrooks EH, Wszolek ZK. Novel Neuroimaging Pattern in POLR3A-Related Disorder on 7T MRI. Neurol Genet. 2024 Jan 10;10(1):e200125. doi: 10.1212/NXG.0000000000200125. eCollection 2024 Feb. No abstract available. PMID 38213753
- [Result] Zaitsu M, Kono K, Hosokawa Y, Miyamoto M, Nanishi K, Okawa S, Niki S, Takahashi K, Yoshihara S, Kobashi G, Tabuchi T. Maternal heated tobacco product use during pregnancy and allergy in offspring. Allergy. 2023 Apr;78(4):1104-1112. doi: 10.1111/all.15536. Epub 2022 Oct 11. PMID 36176042